CLINICAL TRIAL: NCT01027026
Title: The Acute Coronary Syndrome Study. Organization and Treatment of Patients With Acute Coronary Syndrome, With a Focus on Costs, Organization and Security
Brief Title: The Acute Coronary Syndrome Study
Acronym: ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Bilde og Intervensjonsklinikken Radiologi og Nukleaermedisin, Ullevaal University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REK: 6.2008.1724
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Cost analysis; Safety; Length of stay; Randomized controlled trials; Early discharge
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Fast Track Group (Experimental): The patients are discharged the same day after coronary angiography to the refering Hospital
  Interventions: Other: Early discharge
- Group 2: Ordinary care (Active Comparator): Ordinary Cardiology care in the Intervention hospital
  Interventions: Other: Care as usual. No intervention. (Control group)

INTERVENTIONS:
Other: Early discharge — The patients are discharged the same day as coronary angiography.
  Arms: Group 1 Fast Track Group
Other: Care as usual. No intervention. (Control group) — The patients are admitted and cared as usual in cardiology ward.
  Arms: Group 2: Ordinary care

SUMMARY:
The investigators will make a prospective study in which they will look at the economics and security of the treatment of patients with acute coronary syndrome.

The investigators want to do a randomized trial. One group will be treated as they have been treated at Ullevål University Hospital (UUS) in recent years, and the other group will be returned to their refering hospital the same day. The objective of this study will be to provide increased knowledge about whether the rapid discharge from the intervention center is associated with differences in costs or security.

DETAILED DESCRIPTION:
The topic of this study is whether patients with Acute coronary syndrome (ACS)may can be transferred to their refering hospital same day that they arrived intervention hospital.

This is to see if one can reduce the hospital stay and costs for the intervention center, and the total hospitalization time.

and this rapid transport not give more medical complications

Our 1 hypothesis is that patients with ACS, who are transported back to the refering hospital the same day, will reduce the length of stay in intervention center without an increase for the stay at the refering hospital.

Our 2 hypothesis is that patients with ACS, who are transported back to the refering hospital the same day as the treatment is performed, have no more complications than those who stay overnight in the intervention hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients with acute coronary syndrome who are referred from other hospitals

Exclusion Criteria:

* Patients younger than 18years.
* Known mental retardation, dementia or harmful use of alcohol or drugs.
* Allergy or intolerance to ASA and / or clopidogrel.
* Patients who have previously been involved in this study.
* Acute STEMI infarction for less than 72 hours ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-06 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Cost effectiveness. Adverse medical events | 30 days and a year's events

SECONDARY OUTCOMES:
SF-36 | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Ullevaal, Oslo, Norway